CLINICAL TRIAL: NCT06081335
Title: Can Instrumentation Kinematics Affect Post Operative Pain and Substance P Levels? A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Salma Talaat, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 945
Record Dates: First submitted 2023-09-25; First posted 2023-10-13 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Pain, Postoperative; Irreversible Pulpitis; Apical Periodontitis
Keywords: pain; substance P; continuous rotation; reciprocation
MeSH Terms: conditions — Pain, Postoperative; Periapical Periodontitis; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Rotation group (Active Comparator): EdgeEndo x7 continuous rotation files system (Albuquerque, New Mexico, USA)
  Interventions: Device: EdgeEndo x7 continuous rotation files
- Reciprocation group (Active Comparator): EdgeOne Fire reciprocating files system (Albuquerque, New Mexico, USA)
  Interventions: Device: EdgeOne Fire reciprocating files

INTERVENTIONS:
Device: EdgeEndo x7 continuous rotation files — endodontic files operating in continuous rotation
  Arms: Continuous Rotation group
Device: EdgeOne Fire reciprocating files — endodontic files operating in reciprocating motion
  Arms: Reciprocation group

SUMMARY:
The aim of this study was to evaluate the effect of continuous rotation and reciprocation kinematics on post operative pain and difference in substance P levels in patients with irreversible pulpitis with symptomatic apical periodontitis. Twenty patients were randomly distributed into two groups; Continuous Rotation group(n=10): received mechanical preparation using EdgeEndo x7 rotary system (Albuquerque, New Mexico, USA), while Reciprocation group(n=10): received mechanical preparation using EdgeOne Fire reciprocating system (Albuquerque, New Mexico, USA). Apical fluid(AF) samples were collected, and substance P (SP) levels were measured using radioimmunoassay and postoperative pain was measured using Numerical Rating Scale (NRS) preoperatively, at 6h, 12h, 24h, 48h and 72h.

ELIGIBILITY:
Inclusion Criteria:

* Single rooted mandibular second premolar teeth with complete root formation
* Pulpal diagnosis: Symptomatic irreversible pulpitis
* Periapical diagnosis: symptomatic apical periodontitis with no visible periapical radiolucent area
* Patients with pre-operative pain records above 4 on Numerical Rating Scale (NRS) to ensure standardization

Exclusion Criteria:

1. The presence of any systemic disease or allergic reactions
2. Pregnant and lactating females
3. Patients on antibiotic or anti-inflammatory medication
4. Use of analgesics a week prior to treatment
5. A radiographically untraceable canal or an excessively curved root
6. The presence of periapical radiolucency or sinus tract.
7. Teeth with open apices
8. Severe periodontal disease (generalized or localized to the tooth in question)
9. Absence of bleeding in the pulp chamber on access cavity preparation
10. Internal or external resorption

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
difference in substance P levels | pre-operatively and after 5 days at the beginning of the second visit
  tested by radioimmunacy (ELISA)
post operative pain levels | pre-operative, after 6 hours, 12 hours , 24 hours, 48 hours, 72 hours
  Numerical Rating Scale was used to assess pain where 0 is no pain and 10 is the worst possible pain

CONTACTS AND LOCATIONS:
Overall Officials: maram obeid, Study Chair — professor
Locations (2):
- Egypt (2):
  - Ain Shams University, Cairo, Select A State Or Province
  - Ain Shams University, Cairo

REFERENCES:
- [Derived] Abdel-Baset ST, Fahmy SH, Obeid MF. Can instrumentation kinematics affect postoperative pain and substance P levels? A randomized controlled trial. BMC Oral Health. 2024 Jan 17;24(1):102. doi: 10.1186/s12903-024-03882-x. PMID 38233887